CLINICAL TRIAL: NCT06034470
Title: Phase 1 Study of FLAG-Ida With Pivekimab Sunirine (PVEK [IMGN632]) for Adults With Newly Diagnosed Adverse-Risk Acute Myeloid Leukemia and Other High-Grade Myeloid Neoplasms
Brief Title: Combination Chemotherapy (FLAG-Ida) With Pivekimab Sunirine (PVEK [IMGN632]) for the Treatment of Newly Diagnosed Adverse Risk Acute Myeloid Leukemia and Other High-Grade Myeloid Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RG1123378; NCI-2023-03572 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020122 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-08-18; First posted 2023-09-13 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; Mixed Phenotype Acute Leukemia; Myelodysplastic Syndrome; Myelodysplastic/Myeloproliferative Neoplasm; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders | interventions — Specimen Handling; Biopsy; Cytarabine; fludarabine; Granulocyte Colony-Stimulating Factor; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (PVEK, FLAG-Ida) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Procedure: Echocardiography; Drug: Fludarabine; Drug: Granulocyte Colony-Stimulating Factor; Drug: Idarubicin; Procedure: Multigated Acquisition Scan; Drug: Pivekimab Sunirine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspirate
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Granulocyte Colony-Stimulating Factor — Given SC
  Other Names: Colony Stimulating Factor 3; Colony-Stimulating Factor (Granulocyte); Colony-Stimulating Factor 3; CSF3; G CSF; G-CSF; Granulocyte Colony Stimulating Factor; Pluripoietin
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-Demethoxydaunorubicin; 4-DMDR
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Pivekimab Sunirine — Given IV
  Other Names: Anti-CD123 ADC IMGN632; Antibody-drug Conjugate IMGN632; CD123-targeted ADC IMGN632; IMGN 632; IMGN-632; IMGN632

SUMMARY:
This phase I trial finds the best dose of PVEK when given together with fludarabine, cytarabine, granulocyte colony-stimulating factor (G-CSF), and idarubicin, (FLAG-Ida) regimen and studies the effectiveness of this combination therapy in treating patients with newly diagnosed adverse risk acute myeloid leukemia (AML) and other high-grade myeloid neoplasms. PVEK is a monoclonal antibody linked to a chemotherapy drug. PVEK is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as CD123 receptors, and delivers the chemotherapy drug to kill them. Chemotherapy drugs, such as idarubicin, fludarabine, high-dose cytarabine work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. G-CSF helps the bone marrow make more white blood cells in patients with low white blood cell count due to cancer treatment. Giving PVEK with the FLAG-Ida regimen may be a safe and effective treatment for patients with acute myeloid leukemia and other high-grade myeloid neoplasms.

DETAILED DESCRIPTION:
OUTLINE: This is a dose-escalation study of PVEK.

INDUCTION THERAPY: Patients receive PVEK intravenously (IV) on day 1 or day 1 and 22. Patients also receive G-CSF subcutaneously (SC) on days 0-5, fludarabine IV over 30 minutes on days 1-5, cytarabine IV over 2 hours on days 1-5, and idarubicin IV on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients who still have cancer after the first cycle of study treatment may receive an additional cycle of induction chemotherapy with PVEK. Patients who go into remission after the first 1 or 2 cycles of study continue to Post-Remission Therapy.

POST-REMISSION THERAPY: Patients receive PVEK IV on day 1 or day 1 and 22 of each cycle and high-dose cytarabine IV every 12 hours on days 1-6 of each cycle. Treatment repeats every 42 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

Patients also undergo bone marrow aspiration and may undergo bone marrow biopsy and blood sample collection throughout the trial. Patients also undergo echocardiography (ECHO) or multigated acquisition (MUGA) scan during screening and as clinically indicated on trial.

After completion of study treatment, patients are followed every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of untreated AML other than acute promyelocytic leukemia (APL) with t(15;17)(q22;q12) or variants according to the 5th edition of the World Health Organization (WHO) classification of hematolymphoid tumors. Patients with myelodysplastic, myeloproliferative, or myelodysplastic/myeloproliferative neoplasms and ≥ 10% blasts in blood and/or bone marrow, are also eligible, as are patients with mixed phenotype acute leukemia (MPAL). Outside diagnostic material is acceptable to establish diagnosis; submission of peripheral blood specimen for flow cytometry performed at the study institution should be considered. Diagnostic material must have been submitted for cytogenetic and/or molecular testing as clinically appropriate
* Cytogenetically/molecularly adverse-risk disease (European LeukemiaNet [ELN] 2022 criteria)
* Expression of CD123 on immunophenotypically abnormal blasts, as assessed by local multiparameter flow cytometry. Evaluation of CD123 expression via immunohistochemistry is permissible, for example if flow cytometric assessment is not available
* Medically fit, as defined by treatment-related mortality (TRM) score ≤ 13.1 calculated with simplified model
* The use of hydroxyurea prior to start of study therapy is allowed. Patients with symptoms/signs of hyperleukocytosis, white blood cell count (WBC) > 100,000/μL or with concern for other complications of high tumor burden (e.g. disseminated intravascular coagulation) can be treated with leukapheresis prior to start of study therapy
* Patients may have received low-intensity treatment (e.g. azacitidine/decitabine, lenalidomide, growth factors) for antecedent low-grade myeloid neoplasm (i.e. < 10% blasts in blood and bone marrow)
* Bilirubin =< 1.5 x institutional upper limit of normal (IULN) unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x IULN unless elevation is thought to be due to hepatic infiltration by AML
* Creatinine clearance >= 60 mL/min
* Left ventricular ejection fraction >= 45%, assessed by multigated acquisition (MUGA) scan or echocardiography or other appropriate diagnostic modality and no clinical evidence of congestive heart failure
* Fertile male and female subjects must be willing to use an effective contraceptive method before, during, and for at least 3 months after receiving the investigational agent
* Provide written informed consent

Exclusion Criteria:

* Diagnosis of blast phase chronic myeloid leukemia (CML)
* Patients with FLT3-mutated AML
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with antimicrobials, and/or controlled or stable (e.g. if specific, effective therapy is not available/feasible or desired [e.g. known chronic viral hepatitis, human immunodeficiency virus (HIV)]). Patient needs to be clinically stable as defined as being afebrile and hemodynamically stable for 24 hours. Patients with fever thought to be likely secondary to leukemia are eligible
* Known hypersensitivity to any study drug or prior >= grade 3 hypersensitivity reactions to monoclonal antibodies
* Confirmed or suspected pregnancy or active breast feeding
* Treatment with any other investigational anti-leukemia agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities during cycle 1 | During cycle 1 on day 42, or the start of the next cycle
  Dose-limiting toxicities (DLTs) for trial monitoring are defined as follows: a) Any Grade ≥4 organ toxicity; and b) prolonged severe myelosuppression, as defined by ANC <500/µL and platelet count <25,000/µL, for >42 days after initiation (day 1) of FLAG-Ida chemotherapy in the absence of residual disease (assessed by European LeukemiaNet [ELN] response criteria).

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Will be assessed by the NCI CTCAE v.5. Will be analyzed using standard methods for such data: Wilcoxon-rank sum tests for quantitative data; Fisher's exact test for categorical data; Kaplan-Meier, Cox regression, and log-rank tests for time-to-event data.
Measurable residual disease (MRD) rates | Up to 5 years
  Will be estimated within the limits of the study with pivekimab sunirine (PVEK) + fludarabine, high-dose cytarabine, granulocyte colony-stimulating factor, and idarubicin (FLAG-Ida) across study cohorts. Will be analyzed using standard methods for such data: Wilcoxon-rank sum tests for quantitative data; Fisher's exact test for categorical data; Kaplan-Meier, Cox regression, and log-rank tests for time-to-event data.
MRD status | Up to 5 years
  MRD will be measured by multiparameter flow cytometry. All positive testing will be considered positive.
Relapse-free survival | From the date of achievement of remission until the date of hematologic relapse or death from any cause, assessed up to 5 years
  Will be assessed within the limits of the study by the relationship between MRD status after induction therapy and relapse risk/time to relapse. Will be analyzed using standard methods for such data: Wilcoxon-rank sum tests for quantitative data; Fisher's exact test for categorical data; Kaplan-Meier, Cox regression, and log-rank tests for time-to-event data.
Overall survival | From day 1 of study treatment to the date of death from any cause, up to 5 years
  Will be analyzed using standard methods for such data: Wilcoxon-rank sum tests for quantitative data; Fisher's exact test for categorical data; Kaplan-Meier, Cox regression, and log-rank tests for time-to-event data.
Complete remission rates | Up to 5 years
  Will be analyzed using standard methods for such data: Wilcoxon-rank sum tests for quantitative data; Fisher's exact test for categorical data; Kaplan-Meier, Cox regression, and log-rank tests for time-to-event data.
Duration of cytopenias | Up to 5 years
  Will be evaluated by the impact of PVEK dosing regimens on the duration of cytopenias. Will be analyzed using standard methods for such data: Wilcoxon-rank sum tests for quantitative data; Fisher's exact test for categorical data; Kaplan-Meier, Cox regression, and log-rank tests for time-to-event data.
Proportion of patients receiving allogeneic hematopoietic cell transplantation | Up to 5 years
  Will be estimated within the limits of the study by the proportion of patients receiving allogeneic HCT in remission with PVEK + FLAG-Ida. Will be analyzed using standard methods for such data: Wilcoxon-rank sum tests for quantitative data; Fisher's exact test for categorical data; Kaplan-Meier, Cox regression, and log-rank tests for time-to-event data.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Appelbaum, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No